CLINICAL TRIAL: NCT03928587
Title: Effect of 12 Months Supplementation With a Symbiotic Lozenge on Caries Increment in Healthy Children: A Randomized, Parallel-grouped, Placebo-controlled Trial
Brief Title: Effect of 12 Months Supplementation With a Symbiotic Lozenge on Caries Increment in Healthy Children
Acronym: PiP-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-IM-034
Record Dates: First submitted 2019-04-17; First posted 2019-04-26 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): A lozenge containing 2 billion CFU in total of the two strains Lactobacillus paracasei subsp. paracasei and Lactobacillus rhamnosus and arginine 2% to be taken once daily
  Interventions: Dietary Supplement: 2 billion CFU in total of the two strains Lactobacillus paracasei subsp. paracasei and Lactobacillus rhamnosus and arginine.
- Placebo (Placebo Comparator): An identical lozenge except for the absence of probiotics and arginine to be taken once daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 2 billion CFU in total of the two strains Lactobacillus paracasei subsp. paracasei and Lactobacillus rhamnosus and arginine. — One lozenge once daily for 12 months
  Arms: Active
Dietary Supplement: Placebo — Placebo once daily for 12 months
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the effect of a symbiotic lozenge on dental caries in young children.

DETAILED DESCRIPTION:
The study is a multicentre, randomized, double-blind, placebo-controlled, parallel-group study in healthy children aged 5-8 years. The objective is to investigate the effect of a symbiotic lozenge on caries increment in primary molar teeth, primary canines and erupted occlusal surfaces at the first permanent molar teeth.The study will take place in Helsingør and Fredensborg municipality.

The study consists of a baseline visit prior to a 12 months intervention period, followed by a visit after completion. During the intervention period, two to four months after the baseline visit, a saliva sample will be collected.

All guardians to the subjects are encouraged to 1) brush their children's teeth twice daily with the fluoride toothpaste provided, 2) avoid the food provided in appendix D and 3) to continue the subject's dental appointments at local Public Dental Health Service (PDHS). No further specific oral hygiene or dietary instructions/restrictions are provided.

Assuming a dropout rate of 12.5%, 175 children will be included in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children with absence of severe chronic disease
2. Age 5-8 years, both inclusive, at inclusion
3. Ability to cooperate at dental examination
4. Ability to cooperate to a daily intake of a lozenge
5. Parents/legal guarding provided voluntary written informed consent

Exclusion Criteria:

1. Children with severe medical conditions
2. Mentally or physically disabled children
3. Children of parents with language barriers and not able to give written informed consent

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 343 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Increase in caries incidence | 12 months
  Caries increment in primary molar teeth, primary canines and erupted occlusal surfaces at the first permanent molar teeth in children aged 5-8 years, using a modified dmf-s scale, including the occlusal surfaces of the first permanent teeth where d is defined by ICDAS scale and assessed both clinically and by dental x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Azam Bakhshandeh, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porksen CJ, Ekstrand KR, Markvart M, Larsen T, Garrido LE, Bakhshandeh A. The efficacy of combined arginine and probiotics as an add-on to 1450 ppm fluoride toothpaste to prevent and control dental caries in children - A randomized controlled trial. J Dent. 2023 Oct;137:104670. doi: 10.1016/j.jdent.2023.104670. Epub 2023 Aug 20. PMID 37604396
- [Derived] Porksen CJ, Keller MK, Damholt A, Frederiksen AKS, Ekstrand KR, Markvart M, Larsen T, Bakhshandeh A. The effect of a lozenge combining prebiotic arginine and probiotics on caries increment in children during 10-12 months, a randomized clinical trial. J Dent. 2023 Aug;135:104599. doi: 10.1016/j.jdent.2023.104599. Epub 2023 Jun 24. PMID 37356561